CLINICAL TRIAL: NCT00326950
Title: Phase I Clinical Study of E7389 in Patients With Solid Tumors
Brief Title: Phase I Clinical Study of E7389
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-J081-105
Record Dates: First submitted 2006-05-16; First posted 2006-05-17 (Estimated); Results first posted 2011-12-20 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Cancer
Keywords: Cancer; Tumors; Phase I; E7389
MeSH Terms: conditions — Neoplasms | interventions — eribulin

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: E7389

INTERVENTIONS:
Drug: E7389 — E7389 will be administered intravenously on Days 1 and 8 of a 21 day cycle. The initial dose level will be 0.7 mg/m2, with planned dose levels of 1.0, 1.4, 2.0 mg/m2.

SUMMARY:
The primary objective of this study is to determine the dose limiting toxicity and maximum tolerated dose of E7389 in patients with solid tumors. The secondary objectives are to investigate the pharmacokinetics, safety, estimated recommended dose, and anti-tumor effects (in evaluable cases) of E7389 in patients with solid tumors.

ELIGIBILITY:
Inclusion criteria:

1. Patients with histologically or cytologically confirmed solid tumors.
2. Patients who have progressed on or following standard therapy and with no other treatment options.
3. Patients aged 20-74 when they give informed consent.
4. Patients having a performance status (PS) of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
5. Patients who can stay at the hospital from the start of the study drug treatment to 2 weeks of the first cycle.
6. Patients having adequate function of major organs (bone marrow, liver, kidney and lungs):

(1) Neutrophil count 1,500/mm3 (2) Platelet count 100,000/mm3 (3) Hemoglobin 9.0 g/dL (4) Aspartate aminotransferase [AST] 2.5 times the upper limits of normal (ULN) in institute, unless related to liver involvement by tumor, in which case 5.0 times ULN (5) Alanine aminotransferase [ALT] 2.5 times ULN in institute, unless related to liver involvement by tumor, in which case 5.0 times ULN (6) Total bilirubin 1.5 times ULN in institute (7) Serum creatinine 1.5 times ULN in institute (8) Pulse oximeter oxygen saturation 90%

7. Patients with no adverse drug reactions (excluding alopecia, etc.) that were caused by the prior therapy or could influence the safety evaluation of the study drug.

The withdrawal periods required from the completion of the prior therapy to the start of the study drug therapy are as follows:

1. Chemotherapy (excluding oral 5-FU and molecular target drugs), surgical therapy, other study drugs: 4 weeks
2. Nitrosourea agents, mitomycin C: 6 weeks
3. Radiotherapy, endocrinotherapy, immunotherapy, oral 5-FU, molecular target drugs, blood transfusion, blood products, G-CSF and other hematopoietic factors: 2 weeks

8. Patients who give written informed consent.

9. Patients with an expected survival of longer than 3 months from the start of the study drug therapy.

Exclusion criteria:

1. Patients with systemic infection with a fever (38°C).
2. Patients with a large amount of pleural effusion, ascites and pericardial fluid requiring drainage.
3. Patients with brain metastasis with clinical symptoms.
4. Patients with serious complications: (1) Patients with uncontrollable cardiac disease such as ischemic heart disease and arrhythmia at a level of severity that needs to be treated (excluding left ventricular hypertrophy, mild left ventricular volume overload and mild right leg block that accompany hypertension) (2) Patients with myocardial infarction within 6 months prior to study entry (3) Patients with a complication of hepatic cirrhosis (4) Patients with interstitial pneumonia and pulmonary fibrosis (5) Patients with a bleeding tendency
5. Women who are pregnant or breastfeeding, or premenopausal women of childbearing potential.

   Post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Premenopausal women of childbearing potential with either a positive pregnancy test at screening or no pregnancy test, or have not agreed to use adequate measures of contraception.
6. Fertile men who are not willing to use contraception or fertile men with a female partner who is not willing to use contraception.
7. Patients who have tested positive for human immunodeficiency virus (HIV), hepatitis C virus (HCV) antibody, or hepatitis B virus surface antigen (HBsAg).
8. Patients who need continuous systemic steroid therapy during the study period.
9. Patients who need continuous use of phenytoin, carbamazepine, rifampicin and/or barbiturate which induces cytochrome P450 (CYP3A4), a drug-metabolizing enzyme, during the study period.
10. Patients who have received extensive radiation therapy (30% or more of bone marrow).
11. Patients who refused to receive a supportive therapy of blood transfusion by suppressing bone marrow.
12. Patients who are participating in other clinical studies.
13. Patients whom the investigator or subinvestigator has judged inappropriate for this study.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-06; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomio Nakamura, Study Director — Eisai Co., Ltd.
Locations (1):
- Kashiwa, Chiba, Japan

REFERENCES:
- [Derived] Mukohara T, Nagai S, Mukai H, Namiki M, Minami H. Eribulin mesylate in patients with refractory cancers: a Phase I study. Invest New Drugs. 2012 Oct;30(5):1926-33. doi: 10.1007/s10637-011-9741-2. Epub 2011 Sep 2. PMID 21887501

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 1 center in Japan during the period of May 2006 to Jan 2008
Groups:
- E7389: E7389 will be administered intravenously on Days 1 and 8 of a 21-day cycle. Initial dose level will be 0.7 mg/m^2, with planned dose levels of 1.0, 1.4, & 2.0 mg/m^2.
Period: Overall Study
Arm/Group | E7389
Started | 15
Completed | 14
Not Completed | 1
Not completed — Progressive Disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | E7389
Number analyzed (Participants) | 15
Age Continuous [Mean (Standard Deviation); unit: years] | 58.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants] — Subjects were Japanese
  Participants
    American Indian or Alaska Native | 0
    Asian | 15
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Japan | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Experienced Dose Limiting Toxicity (DLT)
Description: DLT is an adverse drug reaction defined as 1)Grade 4 neutropenia for 5 days, 2)>/=Grade 3 febrile neutropenia, 3)>/=Grade 3 neutropenia requiring iv antibiotics, 4)Grade 4 thrombocytopenia, 5)>/=Grade 3 nonhematologic toxicity, 6)Omission of study drug on Day 8 due to >/=Grade 3 neutropenia or thrombocytopenia or investigator decision.
Time Frame: 3 weeks
Measure: Number; unit: participants
Groups:
- E7389: E7389 will be administered intravenously on Days 1 and 8 of a 21 day cycle. The initial dose level will be 0.7 mg/m^2, with planned dose levels of 1.0, 1.4, 2.0 mg/m^2.
Arm/Group | E7389
Number analyzed (Participants) | 15
participants | 5

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD was the lowest dose at which a dose limiting toxicity occurred.
Time Frame: 3 Weeks
Measure: Number; unit: mg/m^2
Arm/Group | E7389
Number analyzed (Participants) | 15
mg/m^2 | 2.0

3. Secondary Outcome: Safety, Tolerability, the Pharmacokinetics, a Recommended Dose (RD) for Phase II Clinical Study and the Anti-tumor Effect in Evaluable Subjects.
Time Frame: 3 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | E7389
Serious Adverse Events (participants affected / at risk) | 5/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E7389 (N=15)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Myelodysplastic Syndrome (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E7389 (N=15)
Febrile Neutropenia (Blood and lymphatic system disorders) | 5
Nasopharyngitis (Infections and infestations) | 2
Pharyngitis (Injury, poisoning and procedural complications) | 1
Pneumonia (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Anorexia (Metabolism and nutrition disorders) | 9
Convulsion (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Neuralgia (Nervous system disorders) | 1
Neuropathy (Nervous system disorders) | 1
Neuropathy Peripheral (Nervous system disorders) | 3
Peripheral Sensory Neuropathy (Nervous system disorders) | 2
Lacrimation Increased (Eye disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Gingivitis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Stomatitis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 8
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Hemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Fatigue (General disorders) | 9
Edema (General disorders) | 3
Edema Peripheral (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 5
Alanine Aminotransferase Increased (Investigations) | 6
Aspartate Aminotransferase Increased (Investigations) | 9
Blood Albumin Decreased (Investigations) | 5
Blood Bilirubin Increased (Investigations) | 1
Blood Calcium Increased (Investigations) | 1
Blood Chloride Increased (Investigations) | 2
Blood Cholesterol Decreased (Investigations) | 1
Blood Cholesterol Increased (Investigations) | 1
Blood Creatine Phophokinase Increased (Investigations) | 4
Blood Creatinine Increased (Investigations) | 1
Blood Glucose Increased (Investigations) | 12
Blood Lactate Dehydrogenase Increased (Investigations) | 3
Blood Potassium Decreased (Investigations) | 2
Blood Sodium Decreased (Investigations) | 3
Blood Urea Decreased (Investigations) | 1
Blood Urea Increased (Investigations) | 1
C-Reactive Protein Increased (Investigations) | 10
Electrocardiogram QT Prolonged (Investigations) | 1
Electrocardiogram ST Segment Depression (Investigations) | 1
Gamma Glutamyltransferase Increased (Investigations) | 5
Glucose Urine Present (Investigations) | 3
Blood Urine Present (Investigations) | 2
Hemoglobin Decreased (Investigations) | 9
Lymphocyte Count Decreased (Investigations) | 13
Neutrophil Count Decreased (Investigations) | 12
Neutrophil Count Increased (Investigations) | 2
Platelet Count Decreased (Investigations) | 5
Protein Total Decreased (Investigations) | 1
Red Blood Cell Count Decreased (Investigations) | 9
Weight Decreased (Investigations) | 1
White Blood Cell Count Decreased (Investigations) | 13
White Blood Cell Count Increased (Investigations) | 2
Protein Urine Present (Investigations) | 4
Blood Alkaline Phosphatase Increased (Investigations) | 3
Tooth Fracture (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No